CLINICAL TRIAL: NCT04373304
Title: The Effect of a Low FODMAP Diet in Irritable Bowel Syndrome Patients
Acronym: FIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, prof.dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s63269
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Irritable Bowel Syndrome; FODMAP
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Masking Description: Patients are blinded during reintroduction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low FODMAP diet (Experimental)
  Interventions: Other: low FODMAP diet

INTERVENTIONS:
Other: low FODMAP diet — A diet specifically developed for the management of IBS is the low Fermentable Oligosaccharides, Disaccharides, Monosaccharides, And Polyols (FODMAP) diet. FODMAP is a collective term that includes fructose in excess of glucose, oligosaccharides including fructans/fructo-oligosaccharides (FOS), galacto-oligosaccharides, sugar polyols such as sorbitol and mannitol, and lactose. Controlled studies have established efficacy of the low FODMAP in managing IBS symptoms, but this diet is complex, associated with low calorie intake, and requires individualized explanation and follow-up by an experienced dietician.

SUMMARY:
Tertiary care IBS patients will be recruited for a prospective low FODMAP intervention study, hereby focusing on the reintroduction phase of the diet, where patients are blindly challenged with different FODMAP groups administered as powder, to be added to the strict FODMAP exclusion phase. During the screening phase of two weeks, baseline data regarding psychological, nutritional, microbial, and genetics will be collected. Predictors of treatment response (a 50-point drop on the IBS-severity scoring system (IBS-SSS) during the strict FODMAP exclusion phase of 6 weeks) will be studied with linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study if all of the following criteria are met:

  1. Patients with irritable bowel syndrome as per Rome IV diagnostic criteria
* Symptom characteristics of IBS according to Rome IV criteria 2. Patients must provide witnessed written informed consent prior to any study procedures being performed 3. Patients aged between 18 and 70 years inclusive 4. Male or female patients

Exclusion Criteria:

* Patients are excluded from the study if any of the following criteria are met:

  1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
  2. Patients with any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years
  3. Patients presenting with predominant symptoms of functional dyspepsia (FD) and of gastro-oesophageal reflux disease (GERD)
  4. Patients who changed their diet over the last 3 months or have previously tried the low FODMAP diet are excluded from the study.
  5. Females who are pregnant or lactating are excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) | approximately 2 years
  The primary endpoint is the variable used to assess the main objective, the efficacy of low FODMAP diet on gastrointestinal symptoms in IBS (focusing on the reintroduction phase). The variables used will be the symptom scores of several symptom questionnaires. Ultimately, the efficacy of the diet is based on improvement of symptom scores. Improvement is defined as a 50-point drop on the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS). In this questionnaire, each quesiton is scored from 0-100, with a maximum total score of 500. Patients reporting scores <50 are defined as non-IBS individuals, a score from 50-175 indicated mild disease, 175-300 moderate and >300 severe.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van den Houte K, Colomier E, Routhiaux K, Marien Z, Schol J, Van den Bergh J, Vanderstappen J, Pauwels N, Joos A, Arts J, Caenepeel P, De Clerck F, Matthys C, Meulemans A, Jones M, Vanuytsel T, Carbone F, Tack J. Efficacy and Findings of a Blinded Randomized Reintroduction Phase for the Low FODMAP Diet in Irritable Bowel Syndrome. Gastroenterology. 2024 Jul;167(2):333-342. doi: 10.1053/j.gastro.2024.02.008. Epub 2024 Feb 23. PMID 38401741